CLINICAL TRIAL: NCT03092180
Title: Optimizing Treatment on Idiopathic Inflammatory Myopathies
Status: Recruiting | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Samuel Katsuyuki Shinjo, PhD, Principal Investigator, University of Sao Paulo
Other Study IDs: MYO-HCFMUSP-01
Record Dates: First submitted 2017-03-09; First posted 2017-03-27 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Idiopathic Inflammatory Myopathies
Keywords: Dermatomyositis; Immunomodulation; Immunosuppressive agents; Myositis; Polymyositis; Necrotizing myopathies; Antisynthetase syndrome
MeSH Terms: conditions — Myositis; Dermatomyositis; Polymyositis; Antisynthetase syndrome | interventions — Infusions, Intravenous; Dosage Forms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and muscle biopsies
  NOTE: This is a observational study. Subjects in the study will receive a routine care that has been established in our Instituition (diagnostic, therapeutic, biospecimen analysis and retention).
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Idiopathic inflammatory myopathies 1: Intravenous infusion with methyprednisolone / human intravenous immunoglobulin at disease onset
  Interventions: Drug: Intravenous Infusion
- Idiopathic inflammatory myopathies 2: Intravenous infusion with methyprednisolone at disease onset
  Interventions: Drug: Intravenous Infusion

INTERVENTIONS:
Drug: Intravenous Infusion — Intravenous infusion of follow medicine at disease onset: methyprednisolone and/or human intravenous immunoglobulin
  Other Names: Medicine

SUMMARY:
As a T2T, our patients with idiopathic inflammatory myopathies will receive pulse therapies with methyprednisolone and/or human intravenous immunoglobulin, or only methyprednisolone at disease onset.

This scheme is an internal routine protocol of our Service.

DETAILED DESCRIPTION:
To compare two groups of patients as described in Brief Summary.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic inflammatory myopathies

Exclusion Criteria:

* Inclusion body myositis, muscular dystrophies, neoplasia-associated myopathies, overlapped myopathies, others myopathies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Idiopathic inflammatory myopathies
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2005-01; Primary Completion 2024-05-06 (Actual); Study Completion 2024-12-04 (Estimated)

PRIMARY OUTCOMES:
Physician Global Activity | Six months
  This partially validated tool measures the global evaluation by the treating physician of the overall disease activity of the patient at the time of assessment using a 10 cm. visual analogue scale and a 5 point Likert scale.
Patient/Parent Global Activity - | Six months
  This partially validated tool measures the global evaluation by the patient, or by the parent if the patient is a minor, of the patient's overall disease activity at the time of assessment using a 10 cm. visual analogue scale.
Manual Muscle Testing | Six months
  This partially validated tool assesses muscle strength using manual muscle testing (MMT). A 0 - 10 point scale is proposed for use. An abbreviated group of 8 proximal, distal, and axial muscles performs similarly to a total of 24 muscle groups, and is also proposed for use for research studies.
Health Assessment Questionnaire | Six months
  Define the health assessement questionnaire. Pontuaction: 0.00-3.00
Muscle Enzymes | Six months
  This partially validated tool measures the serum activities of at least 2 of the 4 muscle-associated enzymes including creatine phosphokinase (CK), the transaminases (ALT, AST), lactate dehydrogenase (LD) and aldolase.
Myositis Disease Activity Assessment Tool | Six months
  After local anesthesia, a cutaneous incision will be made in lateral thigh face. The biopsy will be done using the Bergstrom needle. Histological (hematoxylin and eosin)/immunohistochemical (CD4, CD8, CD68, CD20, C5b-9, MHCI, MHCII, CD31) analysis will be performed in muscle samples (at baseline and after 12 weeks) in all patients (present study)

SECONDARY OUTCOMES:
Side effects to treatment (glucocorticoid, immunosuppressants and/or human intravenous immunoglobulin) | Six months
  Effect of drugs in disease outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Samuel K Shinjo, PhD, Principal Investigator — Universidade de Sao Paulo - Rheumatology Division
Locations (1):
- Samuel Katsuyuki Shinjo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No